CLINICAL TRIAL: NCT00913562
Title: Effect of Rosuvastatin on Endothelial Function in Patients With Diabetes and Glaucoma
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Garhofer, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-040908
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Glaucoma; Diabetes
Keywords: Ocular Physiology; Regional Blood Flow
MeSH Terms: conditions — Glaucoma; Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Patients with diabetes (Active Comparator): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- Patients with glaucoma (Active Comparator): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- Control patients with diabetes (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Control patients with glaucoma (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — one tablet rosuvastatin 10 mg per day for 12 weeks
  Arms: Patients with diabetes; Patients with glaucoma
Drug: Placebo — one tablet a day for 12 weeks
  Arms: Control patients with diabetes; Control patients with glaucoma

SUMMARY:
Endothelial dysfunction can be seen in a variety of vascular related ocular diseases such as glaucoma or diabetic retinopathy. There is accumulating evidence now that statins may at least partially improve endothelial function in several vascular beds, an effect that is probably independent of the lipid lowering effects of the statins.

Consequently, the current study seeks to investigate whether administration of 10 mg rosuvastatin by mouth (p.o.) for 12 weeks can improve the endothelial function in patients with glaucoma and diabetic retinopathy. For this purpose, flow mediated vasodilatation of the brachial artery and flicker induced vasodilatation of retinal vessels will be measured at baseline, after 6 and 12 weeks of treatment with rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

Diabetes patients:

* Men and women aged over 18 years.
* subjects with both hypercholesterolemia and normal lipid profile will be included.
* Diabetes type I or type II. Only patients with no signs of diabetic retinopathy (level 1) or patients with mild or moderate diabetic retinopathy will be included. Level of diabetic retinopathy will be assessed according to the modified Airlie House classification (1991).
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant.
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant.
* -Normal ophthalmic findings, except diabetic retinopathy as described above, ametropia < 6 Dpt.

Glaucoma patients:

* Men and women aged over 18 years.
* Subjects with both hypercholesterolemia and normal lipid profile will be included.
* Open angle glaucoma defined as pathological optic disc appearance and characteristic visual field loss. Visual field loss is defined as having a glaucoma hemifield test outside normal limits and/or a CPSD with P < 0.05 (Keltner et al. 2003).
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant.
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant.
* Normal ophthalmic findings, except glaucoma as described above, ametropia < 6 Dpt.
* sufficiently controlled intraocular pressure.

Exclusion Criteria:

* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study.
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day.
* Previous or current treatment with statins.
* Current treatment with fibrates.
* History or presence of renal failure, creatine kinase (CK) and lactic dehydrogenase (LDH) above normal levels.
* History or presence of hepatic dysfunction, including increase of liver enzymes.
* Patients with known hypersensitivity to the study drug or any ingredients.
* Patients with or with a history of myopathy.
* Systemic treatment with oral anticoagulants except low dose aspirin.
* Blood donation during the previous 3 weeks.
* Ametropia of 6 or more than 6 dpt.
* Presence of intraocular pathology other than non proliferative diabetic retinopathy for cohort I and glaucoma for cohort II.
* Ophthalmological surgery (including argon laser trabeculoplasty (ALT), trabeculectomy, deep sclerectomy) within the last 6 months before the study.
* History or family history of epilepsy.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Flicker induced vasodilatation | 10 minutes blood flow measurements on 3 study days - up to12 weeks of treatment with rosuvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhofer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria